CLINICAL TRIAL: NCT00230139
Title: The Added Value of SPECT/CT in the Evaluation of Endocrine and Neuroendocrine Tumors
Brief Title: SPECT/CT in Endocrine and Neuroendocrine Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Rambam Health Care Campus, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: endocrineCTIL
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2005-09

CONDITIONS: Endocrine and Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Single Photon Emission Computed Tomography Computed Tomography

INTERVENTIONS:
Device: SPECT/CT

SUMMARY:
The value of fusion of functional and anatomical data has been described using several fusion techniques for various nuclear medicine procedures and morphologic imaging modalities (SPECT-CT, SPECT-MRI, Coincidence-CT). We hypothesize that NM -CT data has advantages over the data obtained using separately performed NM study and conventional anatomic imaging as CT. We hypothesize that more accurate localization of the radio-isotope activity on NM images will improve diagnostic accuracy and will have an impact on patient management:

Improved accuracy of NM study will improve tumor localization, the evaluation of the extent of disease and the post therapy follow up.

It will direct other diagnostic procedures to lesions otherwise undetected, or exclude the need for more invasive procedures. It can also guide invasive procedures and radiation-therapy planning, thus improving therapy results and avoiding unnecessary treatment-related side effects.

DETAILED DESCRIPTION:
The value of fusion of functional and anatomical data has been described using several fusion techniques for various nuclear medicine procedures and morphologic imaging modalities (SPECT-CT, SPECT-MRI, Coincidence-CT). We hypothesize that NM -CT data has advantages over the data obtained using separately performed NM study and conventional anatomic imaging as CT. We hypothesize that more accurate localization of the radio-isotope activity on NM images will improve diagnostic accuracy and will have an impact on patient management:

Improved accuracy of NM study will improve tumor localization, the evaluation of the extent of disease and the post therapy follow up.

It will direct other diagnostic procedures to lesions otherwise undetected, or exclude the need for more invasive procedures. It can also guide invasive procedures and radiation-therapy planning, thus improving therapy results and avoiding unnecessary treatment-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for NM scintigraphy to assess the presence of endocrine or neuroendocrine tumors.
* Patient signed informed consent

Exclusion Criteria:

* The study will not be performed in pregnant or lactating women.
* Patient will not be able or willing to tolerate the scan until its completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2002-01; Primary Completion 2004-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The impact of imaging modality on patient management

SECONDARY OUTCOMES:
The impact of imaging modality on patient management

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Keidar, MD,PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel